CLINICAL TRIAL: NCT04943562
Title: Evaluation of the Viability of Actigraphy, Wearable EEG Band and Smartphone for Sleep Staging in Comparison With Polysomnography
Brief Title: Actigraphy, Wearable EEG Band and Smartphone for Sleep Staging
Status: Recruiting | Type: Observational
Sponsor: SleepUp Tecnologia em Saúde Ltda (Industry)
Responsible Party: Sponsor
Other Study IDs: SleepUp_#02
Record Dates: First submitted 2021-06-13; First posted 2021-06-29 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Sleep; Insomnia; Sleep Apnea Syndrome, Obstructive
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Healthy participants: Participants from 20 to 80 years old, from both genders and with no sleep disorders
  Interventions: Diagnostic Test: ACT+EEG
- Participants with sleep disorders: Participants between the ages of 20 and 80 years who reported one or more sleep-related disorders or complaints. Among these, at least 30% of the sample should have moderate to severe insomnia (as measured by the insomnia severity index), 30% should have high risk to sleep apnea (as measured by the STOP-BANG questionnaire) and 70% should have excessive sleepiness scale (as measured by the Epworth sleepiness scale).
  Interventions: Diagnostic Test: ACT+EEG

INTERVENTIONS:
Diagnostic Test: ACT+EEG — Combination of ACT+EEG. This is not an intervention, but rather a combination of devices to be tested regarding its diagnostic validity.

SUMMARY:
This study aims to evaluate the viability of the combined use of wearable and portable technologies for sleep staging. The results will be compared with polysomnography, in order to achieve clinical and diagnostic validation. Three domains of devices will be used: Movement sensors, wearable EEG band and smartphones

The project will be composed of two stages:

In the first stage, the use of the combination of actigraphy and EEG will be used for sleep staging in a sample of 12 healthy volunteers from 20 to 80 years old, both genders and with no sleep disorders for each combination of ACT+EEG. Considering there will two of each (thus four combinations), the final sample will be composed of 48 individuals. Once recruited, evaluated according to the inclusion and exclusion criteria and consented with the terms of this study, the participants will be referred to the sleep lab, in which they will undergo a full night type-1 in lab polysomnography, following the setup recommended by the American Academy of Sleep Medicine. Concomitantly with the polysomnography, the participants will also use the combination of ACT+EEG.

In the second stage, the most successful combination tested in the first stage will be tested in a clinical sample, composed by 60 participants from both genders, from 20 to 80 years old and with at least one sleep disorder or complaint. Among these, at least 30% of the sample should have moderate to severe insomnia, 30% should have high risk to sleep apnea and 70% should have excessive sleepiness scale. All the procedures, including the polysomnography will be performed identically to the first step.

DETAILED DESCRIPTION:
This study aims to evaluate the viability of the combined use of wearable and portable technologies for sleep staging. The results will be compared with polysomnography, in order to achieve clinical and diagnostic validation. Three domains of devices will be used:

* Movement sensors: Devices equipped with movement sensors (such as an accelerometer) able to monitor movement over the using period, converting this information in data related to the sleep-wakefulness cycle. In this category, the reference devices are the actimeters/actigraphs (ACT). Its use is recommended by the American Academy of Sleep Medicine to the diagnosis of insomnia and circadian sleep disorders, and should be used for 3 to 14 consecutive days. Other wearable devices, such as smartwatches, are also used with the same purpose, although not validated for clinical use. In this study two wearable devices with movement sensors will be used, with the following minimal specifications: accelerometer in three axes, minimal sampling rate of 25Hz, maximum weight of 100g, battery lasting at least a week and support for Bluetooth connection. The desirable criteria are: light, body temperature and hearth rhythm sensors.
* Wearable EEG band: EEG is a mandatory feature for type-1 polysomnography and a requirement for regular sleep staging. In this project, the EEG will be used in combination with actigraphy to allow a better estimation of sleep stages. In this study two wearable EEG bands will be tested, with the following minimal specifications: dry EEG electrode (no need of paste, gel or other conductor), presented as a head band or stripe, minimal sampling rate of 500Hz, noise, high and low filters, battery lasting at least 8h, maximum weight of 200g (including the whole device) and support for Bluetooth connection.
* Smartphones: Additionally to the movement sensors and the EEG bands, the evaluation of sleep pattern will be based on smartphone-based accelerometers. This is the most common approach among the currently available sleep tracking applications, although is the least accurate. In this project the smartphones will be equipped with SleepUp's app and its sleep tracking functionality.

The project will be composed of three stages:

In the first stage, the use of the combination of actigraphy and EEG will be used for sleep staging in a sample of 12 healthy volunteers from 20 to 80 years old, both genders and with no sleep disorders for each combination of ACT+EEG. Considering there will two of each (thus four combinations), the final sample will be composed of 48 individuals. Once recruited, evaluated according to the inclusion and exclusion criteria and consented with the terms of this study, the participants will be referred to the sleep lab, in which they will undergo a full night type-1 in lab polysomnography, following the setup recommended by the American Academy of Sleep Medicine. Concomitantly with the polysomnography, the participants will also use the combination of ACT+EEG.

In the second stage, the most successful combination tested in the first stage will be tested in a clinical sample, composed by 60 participants from both genders, from 20 to 80 years old and with at least one sleep disorder or complaint. Among these, at least 30% of the sample should have moderate to severe insomnia (as measured by the insomnia severity index), 30% should have high risk to sleep apnea (as measured by the STOP-BANG questionnaire) and 70% should have excessive sleepiness scale (as measured by the Epworth sleepiness scale). All the procedures, including the polysomnography will be performed identically to the first step.

ELIGIBILITY:
FIRST STAGE (Healthy volunteers)

Inclusion Criteria:

* Age between 20 and 80 years old
* Living in the city of São Paulo, Brazil
* No physical or intellectual disability that prevent attending to a in-lab polysomnography or understanding its instructions.

Exclusion Criteria:

* Excessive daytime sleepiness (as measured by the Epworth Sleepiness Scale)
* Poor sleep quality (as measured by the Pittsburgh Sleep Quality Index)
* Insomnia symptoms at any level (as measured by the Insomnia Severity Index)
* Symptoms of depression (as measured by the Beck Depression Inventory)
* High risk to sleep apnea (as measured by the Stop-Bang questionnaire)
* Presence of sleep-related symptoms (as measured by the UNIFESP (Federal University of São Paulo sleep questionnaire)
* Self-reported abuse of alcohol, use of abuse drugs or use of medicine that might impact the normal sleep pattern (including hypnotics, benzodiazepines, antidepressants, corticosteroids, etc).
* Self-reported chronic diseases
* Diagnosis of any sleep disorders during the polysomnography

SECONDS STAGE (volunteers with sleep disorders or complaints)

Inclusion Criteria:

* Age between 20 and 80 years old
* Living in the city of São Paulo, Brazil
* No physical or intellectual disability that prevent attending to a in-lab polysomnography or understanding its instructions.
* At least one sleep disorder or sleep complaint. . Among these, at least 30% of the sample should have moderate to severe insomnia (as measured by the insomnia severity index), 30% should have high risk to sleep apnea (as measured by the STOP-BANG questionnaire) and 70% should have excessive sleepiness scale (as measured by the Epworth sleepiness scale).

Exclusion criteria:

* Absence of sleep disorders.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals from both genders, from 20 to 80 years old, healthy (at stage 1) or with at least one sleep disoder or complaint (at stage 2).
Sampling Method: Non-Probability Sample
Enrollment: 96 (Estimated)
Dates: Start 2021-09-09 (Actual); Primary Completion 2021-12-12 (Actual); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Sleep Latency | Immediately after the polysomnography.
  Time from the beginning of the polysomnographic record until the first epoch of sleep.
Total sleep time | Immediately after the polysomnography.
  Total time of epochs staged as sleep.
Sleep efficiency | Immediately after the polysomnography.
  Percentage of sleep in relation to total record/bed time.
Wake after sleep onset | Immediately after the polysomnography.
  Total time of epochs staged as "wake" after sleep latency.
Latency to REM sleep | Immediately after the polysomnography.
  Time from sleep latency until the first epoch of REM sleep.
Total time for each sleep stage | Immediately after the polysomnography.
  Time corresponding to epochs staged as each of the sleep stages (N1, N2, N3 and REM)
Percentage each sleep stage | Immediately after the polysomnography.
  Percentage corresponding to epochs staged as each of the sleep stages (N1, N2, N3 and REM), in comparison with total sleep time.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Pires, PhD, Principal Investigator — Instituto do Sono
Locations (2):
- Brazil (2):
  - SleepUp Tecnologia em Saúde LTDA, São Caetano do Sul, São Paulo
  - Centro de Especialistas do Sono, São Paulo

IPD SHARING:
Plan to Share IPD: No
The dissemination of Individual Participant Data (IPD) from this study is strictly limited by restrictions on the release of intellectual property, concerns regarding participant privacy and confidentiality, and the absence of explicit consent for extensive data sharing. However, upon reasonable request and subject to approval by the study's principal investigator, anonymized datasets may be provided to qualified researchers. It is imperative that requests include a thorough research proposal and a rationale that substantiates the need for the resources in question.

REFERENCES:
- [Derived] Melo MC, da Silva Vallim JR, Garbuio S, Soster LA, Sousa KMM, Bonaldi RR, Pires GN. Validation of a sleep staging classification model for healthy adults based on two combinations of a single-channel EEG headband and wrist actigraphy. J Clin Sleep Med. 2024 Jun 1;20(6):983-990. doi: 10.5664/jcsm.11082. PMID 38427322